CLINICAL TRIAL: NCT03151785
Title: The School Lifesavers Study: A Randomised Controlled Trial Comparing the Impact of Lifesaver Programme Only, Lifesaver With Face-to-face Training and Face-to-face Training Only on CPR Knowledge, Skills and Attitudes in School Children
Brief Title: The School Lifesavers Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Heart of England NHS Trust (Other); Resuscitation Council UK (Unknown); Calderdale and Huddersfield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UoB
Record Dates: First submitted 2016-06-29; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Arrest
Keywords: CPR; Schools; Education; Lifesaver
MeSH Terms: conditions — Heart Arrest

ARMS (3):
- Face-to-face BLS training (Active Comparator): Pupils will receive CPR training by standardised face-to-face BLS training only
  Interventions: Other: Face-to-face BLS training
- Lifesaver training (Active Comparator): Pupils will receive CPR training by Lifesaver programme only
  Interventions: Other: Lifesaver training
- Lifesaver and Face-to-Face BLS training (Active Comparator): Pupils will receive CPR training by Lifesaver and standardised face-to-face BLS training
  Interventions: Other: Lifesaver and Face-to-Face BLS training

INTERVENTIONS:
Other: Face-to-face BLS training — Pupils will receive CPR training by standardised face-to-face BLS training only
  Arms: Face-to-face BLS training
Other: Lifesaver training — Pupils will receive CPR training by Lifesaver programme only
  Arms: Lifesaver training
Other: Lifesaver and Face-to-Face BLS training — Pupils will receive CPR training by Lifesaver and standardised face-to-face BLS training
  Arms: Lifesaver and Face-to-Face BLS training

SUMMARY:
60,000 people suffer an out of hospital cardiac arrest in the United Kingdom (UK) every year. Bystander cardiopulmonary resuscitation (CPR) rates are dismal (30%) compared with places where CPR education is mandatory for all school children (>50%). Strategies are needed to increase these rates through innovative approaches. Lifesaver (www.life-saver.org.uk) is an immersive interactive programme/application that presents such an opportunity. This study aims to assess the effectiveness of Lifesaver on CPR attitudes, knowledge, skills acquisition and retention in school children. Additionally, it aims to examine whether Lifesaver provides additional benefits in terms of CPR attitudes, knowledge, skills acquisitions and retention in school children when combined with face-to-face BLS training.

DETAILED DESCRIPTION:
The UK has one of the highest rates of cardiovascular disease in the world and approximately 60,000 out-of-hospital cardiac arrests occur every year, half of which are attended to by the emergency services. The public health implications of this are significant as the number of out of hospital cardiac arrests will increase with the rising incidence of obesity and other co-morbidities in the UK's ageing population. Basic Life Support (BLS) can improve the outcomes of these people if it is swiftly performed at the scene of the cardiac arrest.

BLS is defined as a set of skills that can be used to 'help keep someone alive in an emergency...before professional help arrives'. One of the main elements of BLS is cardio- pulmonary resuscitation (CPR). Bystander CPR is important because it slows down the rapid decline in a patient's chances of survival while waiting for professional help. If a patient is found to be in a 'shockable rhythm' such as ventricular fibrillation (VF) or ventricular tachycardia (VT) then receiving bystander CPR could treble the chances of survival.

Currently the average bystander CPR rate in the UK is 30%. This figure is very poor when compared to Seattle where the bystander CPR rates are 61% after routinely training school children for the past 32 years. Similar results have also been achieved in Norway.

While educating the lay public in BLS is key to increasing survival from cardiac arrests, it is difficult to reach the entire population. One potential strategy is to educate school children as young as 12 years old. The American Heart Association advocated compulsory resuscitation training in American schools in 2011, and countries in which resuscitation has been integrated into educational programs in schools report significantly higher resuscitation rates. In Denmark, successful training of school children has led to the rate of bystander CPR doubling after 5 years with a threefold improvement in survival following out-of-hospital cardiac arrest over 10 years. A threefold improvement in survival cannot be achieved solely by improvements in professional medical care in this area.

CPR training in school children has many potential benefits. School children at a young age have a less inhibited approach to resuscitation training and both medical professionals and teachers achieve success after appropriate training themselves. The response to instruction is easier and better at a younger age. Research has shown that the strongest factor preventing laypeople to help in real-life cardiac arrest is a fear of making mistakes. This fear can hopefully be prevented when taught during a young age at school. A more favourable attitude to learning is also reflected by the fact that practical training can be communicated in a more positive way. Embedding resuscitation in related school subjects such as biology, sports or health education is possible and it can make it meaningful.

If school children receive such training, they are also likely to teach this to their family at home. Not only will there be an increase in the number of cardiac arrest survivors worldwide, but also the social benefits of enthusiastic and positive young people. They learn to help others and a sense of responsibility can be instilled in children from a young age. School children and teachers are important "multipliers" in both private and public settings and thus, in the longer term, the proportion of trained individuals in society will markedly increase, leading to an increase in the overall rate of lay resuscitation. By teaching school children, CPR training can reach all groups of society including those in lower social groups. To achieve a statistically significant increase in the resuscitation results, it has been estimated that at least 15% of a population need to be trained and such numbers cannot be achieved by offering voluntary courses.

In their systematic review Plant and Taylor found that training school children in CPR from the age of 10 years old is effective. Young children can learn about certain elements of first aid such as the recovery position and making a 999 call which they are able to retain. It has also been shown that early training helps reduces anxieties about making mistakes in an emergency situation and also markedly increases participants willingness to help. Individuals who have received CPR training are more likely to perform bystander CPR than people without training.

In March 2013, the Department of Health published a Cardiovascular Disease Outcomes Strategy. One of their targeted outcomes is "to consider ways of increasing the numbers trained in CPR and using automated external defibrillators (AED)". Delivering BLS training to every school child would achieve this outcome. Using secondary schools to teach first aid would capture a large proportion of the population as it is compulsory to attend secondary education up until 16 years of age. There is a growing level of support for this approach from Health Care Professionals such as Cardiologists. A joint statement was released by the European Patient Safety Foundation (EuPSF), the European Resuscitation Council (ERC), the International Liaison Committee on Resuscitation (ILCOR) and the World Federation of Societies of Anesthesiologists (WFSA) to call for all children across the world to be trained in the performance of CPR. This initiative supports the training of children at the age of 12 for 2 hours per year in emergency life support and has received strong backing from the World Health Organisation.

The investigators literature review revealed learning technology such as computer or multi-media based resuscitation training programs has been previously evaluated. Studies have found that computer- based simulation provided a learning environment with realistic scenarios when compared to traditional classroom-based teaching. Students who participated in computer or multi-media CPR training had equivalent or superior knowledge and skill acquisition when compared with traditional training. Studies that examined the use of new learning technology merely as a vehicle of delivering the same learning content have failed to improve learning. The systematic review by Plant and Taylor concluded that CPR training in school children could be successful using a variety of approaches. In order to engage and capture the attention the current generation of school children, innovative interactive games could be used in CPR training. To date there has been no studies that investigated the use of immersive interactive scenario training as a standalone education tool or in combination with face-to-face instructor-led training.

The investigators believe that Lifesaver Programme can provide age-appropriate training to schoolchildren. The novel 'game-in-film' format of Lifesaver is an immersive interactive website or application which provides an engaging learning experience and real life scenarios whereby the user helps a victim of cardiac arrest of choking. It is free to use and has currently been downloaded over 46,800 times and the website has been visited over 423,000 times. There is already anecdotal evidence of two lives saved as a result. Furthermore, Lifesaver has won a Webby award, five e-Learning Age awards, and was shortlisted for a British Academy of Film and Television Arts (BAFTA) award.

This study aims to assess the effectiveness of Lifesaver on CPR attitudes, knowledge, skills acquisition and retention in school children. Additionally, it aims to examine whether Lifesaver provides additional benefits in terms of CPR attitudes, knowledge, skills acquisitions and retention in school children when combined with face-to-face BLS training.

Three secondary schools in the West Midlands will participate. Parents of the participating school pupils will be provided with detailed and sufficient information to allow them to consent on behalf of their child for participation in the study. After the initial intervention, 2 and 4 month follow up visits will be conducted to assess the retention of the pupils CPR knowledge, skills and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* All secondary schools in West Midlands
* Year 8 pupils

Exclusion Criteria:

* Participation in British Heart Foundation Heartstart programme
* Schools with established CPR training programme for Year 8 and unable to substitute their programme with teaching provided by this study
* Inability to participate in study during allocated timeframe

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Chest compression depth (mm) from day of intervention and at 2 month and 4 month follow up visits. | Day 0, 2 month, 4 month
Change in Chest compression rate from day of intervention and at 2 month and 4 month follow up visits | Day 0, 2 month, 4 month

SECONDARY OUTCOMES:
Change in CPR attitude measured using an attitudes table questionnaire from baseline to post teaching and testing on Day 0 of intervention and at follow up | Baseline on Day 0, Post intervention on Day 0 of testing, 2 month, 4 month
CPR knowledge test using a questionnaire | Post intervention on Day 0 of testing, 2 month, 4 month

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Yeung, Principal Investigator — University of Birmingham